CLINICAL TRIAL: NCT05346146
Title: A Prospective, Single-arm, Exploratory Clinical Study of Sintilimab Injection in Combination With Paclitaxel (Albumin-bound) and Gemcitabine in Translational Therapy in Patients With Unresectable Locally Advanced Pancreatic Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2020-160; ChiCTR2100046345 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Unresectable Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — sintilimab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sintilimab; Gemcitabine; Albumin-paclitaxel — Sintilimab: 200mg IV Q3W D1; Gemcitabine: 1000mg/m2 IV Q3W D1,8; Albumin-paclitaxel：125mg/m2,IV,D1,D8,Q3W

SUMMARY:
Pancreatic cancer is a common malignant tumor of digestive tract, and its morbidity and mortality are increasing worldwide. Few clinical data have been published on immunotherapy for pancreatic cancer. This trial is a prospective, single-arm, single-center clinical study to investigate the efficacy and safety of sintilimab in combination with gemcitabine and albumin-paclitaxel conversion therapy with unresectable locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center clinical study to investigate the efficacy and safety of sintilimab in combination with gemcitabine and albumin-paclitaxel conversion therapy with unresectable locally advanced pancreatic cancer.

The primary endpoint is R0-surgery resection rate. Objective response rate, overall survival , progression-free survival, event free survival, adverse events will be recorded and analyzed, to assess the efficacy and safety of the combination treatment with sintilimab and paclitaxel (albumin-bound) and gemcitabine with metastatic pancreatic cancer. The study will also explore biomarkers that can predict efficacy, and blood and tumor samples will be collected/collected at baseline and during the trial for patients who sign informed consent, including possible tumor biopsies at baseline.

ELIGIBILITY:
Inclusion Criteria:

-

1. Signed the Informed Consent Form; 2. Age ≥18 and ≤ 75, no gender limitation; 3. Histopathological diagnosis of pancreatic cancer; 4. Patients with unresectable initial local progression and no prior antitumor therapy (radiotherapy, chemotherapy, targeted or immunotherapy, etc.); 5. According to the efficacy evaluation criteria for solid tumors (RECIST version 1.1), at least one lesion can be measured on imaging; 6. ECOG score 0-1; 7. Expected survival time >3 months; 8. Adequate organ function, patient shall meet the following laboratory criteria:

1. Absolute value of neutrophils (ANC) ≥1.5x109/L without the use of granulocyte colony-stimulating factor in the last 14 days.
2. Platelets ≥75×109/L in the last 14 days without blood transfusion.
3. Hemoglobin >9g/dL in the absence of blood transfusion or erythropoietin in the last 14 days;
4. total bilirubin ≤2× upper limit of normal value (ULN) or ≤50umol/L;
5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤5×ULN;
6. Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60 mL /min;
7. Good coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN;
8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, patients with total T3 (or FT3) and FT4 within the normal range may be enrolled; 9. For female patients of reproductive age, a negative urine or serum pregnancy test should be performed within 3 days prior to receiving the first study drug administration (day 1 of cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. Women of childbearing age were defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy; 10. If there is a risk of conception, all patients (both men and women) will be required to use a contraceptive with an annual failure rate of less than 1% for the entire treatment period up to 120 days after the last study drug (or 180 days after the last chemotherapeutic drug).

Exclusion Criteria:

* 1. Malignant diseases other than pancreatic cancer were diagnosed within 5 years prior to first administration (excluding radical basal cell carcinoma of the skin, squamous carcinoma of the skin, and/or radical resected carcinoma in situ); 2. Patients who are currently participating in an interventional clinical study or have been treated with another study drug or study device within 4 weeks prior to initial administration; 3. Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibiting T-cell receptor (e.g., CTLA-4, OX-40, CD137); 4. Received systemic therapy with anti-tumor indications of Proprietary Chinese medicines or immunomodulatory drugs (including interferon and interleukin, except local use for ascites control) within 2 weeks before the first administration; 5. An active autoimmune disease requiring systemic therapy (e.g., palliative drugs, glucocorticoids or immunosuppressants) has occurred within 2 years prior to first dosing. Alternative therapies (e.g. thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary dysfunction) are not considered systemic; 6. Patients who were receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation, or other topical glucocorticoid) or any other form of immunosuppressive therapy within 7 days prior to initial dosing; Note: Physiological doses of glucocorticoids (≤10 mg/ day of prednisone or equivalent) are permitted; 7. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation is known; 8. Those who are known to be allergic to active ingredients or excipients of sintilimab, gemcitabine and albumin-paclitaxel; 9. Has not fully recovered from toxicity and/or complications associated with any intervention prior to initiation of treatment (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss); 10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 11. Uncontrolled active hepatitis B (defined as HBsAg positive with hbV-DNA copy number greater than the upper limit of the normal value in the laboratory department of the research center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load <1000 copies/mL (200 IU/ml) before initial administration, subjects should receive anti-HBV therapy throughout study drug therapy to avoid virus reactivation
2. For subjects resistant to HBc (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of virus reactivation is required 12. Active HCV-infected subjects (HCV antibody positive and HCV-RNA level above the detection limit); 13. Received live vaccine within 30 days prior to initial administration (cycle 1, day 1); Note: Acceptance of injectable inactivated virus vaccine against seasonal influenza is permitted within 30 days prior to first administration; Intranasally administered live attenuated flu vaccines are not allowed.

14. Pregnant or lactating women; 15. Presence of any serious or uncontrollable systemic illness, such as:

1. Serious and uncontrollable abnormalities in the rhythm, conduction or morphology of resting electrocardiogram, such as complete left bundle branch block, heart block above degree ⅱ, ventricular arrhythmia or atrial fibrillation;
2. Unstable angina pectoris, congestive heart failure, NYHA grade ≥ 2 chronic heart failure;
3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months prior to treatment inclusion;
4. Poor blood pressure control (systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg);
5. A history of non-infectious pneumonia requiring glucocorticoid treatment within 1 year prior to initial administration, or the current presence of clinically active interstitial lung disease;
6. Active tuberculosis;
7. The presence of active or uncontrolled infections requiring systemic treatment;
8. Clinical active diverticulitis, abdominal abscess and gastrointestinal obstruction;
9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. Poor control of diabetes (FBG > 10mmol/L);
11. Urine routine showed urine protein ≥++, and confirmed 24-hour urine protein quantity > 1.0g;
12. Those with mental disorders and unable to cooperate with treatment; 16. Any medical history or disease evidence that may interfere with the results of the study, abnormal values of treatment or laboratory tests, or other conditions that the researcher considers unsuitable for the study because of other potential risks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
R0-surgery resection rate | up to approximately 12 months
  participants with R0-surgery resection/ all operated patients

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 12 months
Overall survival (OS) | 14 weeks after the initiation of the treatment
Progression Free Survival (PFS) | Up to approximately 12 months
event free survival (EFS) | Up to approximately 12 months
All the adverse events by NCI CTCAE v 5.0 | 12 months

OTHER OUTCOMES:
Biomarkers predictive of response and toxicity | Up to 1 year after start of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided